CLINICAL TRIAL: NCT02404051
Title: Fulvestrant Followed by Everolimus Plus Exemestane vs Examestane and Everolimus Followed by Fulvestrant in Postmenopausal Women With HR+ and HER2- Locally Advanced (LABC) or Metastatic Breast Cancer (MBC) Previously Treated With NSAI
Brief Title: Fulvestrant and EVerolimus Plus EXemestane in Metastatic Breast Cancer
Acronym: FEVEX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorzio Oncotech (Other)
Collaborators: Clinical Research Technology S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIM16-FEVEX; 2014-004035-38 (EudraCT Number)
Record Dates: First submitted 2015-01-26; First posted 2015-03-31 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Metastatic Breast Cancer; Breast Cancer; Hormone Receptor Positive Tumor; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast; Locally Advanced Malignant Neoplasm
Keywords: Breast cancer; HER2Negative; hormone receptor positive (HR+); Metastatic; Locally Advanced; fulvestrant; everolimus; exemestane
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Everolimus; exemestane; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM 1 (Experimental): Everolimus plus Exemestane -> progression disease (PD) -> fulvestrant (ARM 1)
  Interventions: Drug: Everolimus; Drug: Exemestane; Drug: Fulvestrant
- ARM 2 (Experimental): Fulvestrant -> progression disease (PD) -> everolimus plus exemestane (ARM 2)
  Interventions: Drug: Everolimus; Drug: Exemestane; Drug: Fulvestrant

INTERVENTIONS:
Drug: Everolimus — 10 mg daily tablets
  Other Names: Afinitor
Drug: Exemestane — 25 mg daily tablets
  Other Names: Aromasin
Drug: Fulvestrant — 500 mg i.m. on Days 1, 15 and 29 and every 28 days thereafter
  Other Names: Faslodex

SUMMARY:
This is a multi-center, randomized, open-label, parallel group study designed to evaluate efficacy and safety of fulvestrant followed, at progression, by examestane and everolimus versus examestane and everolimus followed, at progression, by fulvestrant in postmenopausal women with HR+ and HER2- LABC or MBC whose disease has progressed to NSAI in the adjuvant or metastatic setting.

DETAILED DESCRIPTION:
In this study everolimus will be administered in combination with exemestane, which is an irreversible steroidal aromatase inactivator that has demonstrated efficacy in the treatment of postmenopausal patients with ABC. Exemestane is indicated for adjuvant treatment of postmenopausal women with HR+ EBC who have received two to three years of tamoxifen and are switched to exemestane for completion of a total of five consecutive years of adjuvant hormonal therapy. It is also indicated for the treatment of ABC in postmenopausal women whose disease has progressed following tamoxifen therapy (in the USA) or following antiestrogen therapy (in Europe). In 2011, the BOLERO-2 trial reported (5; 33) a significant benefit for HR+ HER2- postmenopausal pretreated women in the ABC setting by combining everolimus with exemestane. In this randomized, double-blind, placebo-controlled trial a statistically significant improvement in PFS by adding everolimus to exemestane versus exemestane alone was reported. Adding everolimus determined a 2.4-fold prolongation in PFS from 3.2 up to 7.4 months and so lowered the risk of cancer progression by 56% for these women. These findings were confirmed by an independent assessment (4.1 vs. 11.0 months, risk reduction: 64%). The QoL data shows positive trend in the everolimus plus exemestane treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women (≥ 18 years of age) with LABC or MBC not amenable to curative treatment by surgery or radiotherapy, refractory to NSAI
2. Histological or cytological confirmation of ER+ BC and/or PgR+.
3. Postmenopausal women.
4. Radiological or objective evidence of recurrence or progression on or after the last systemic therapy prior to randomization
5. Patients must have:

   * At least one lesion that can be accurately measured in at least one dimension ≥ 20 mm with conventional imaging techniques or ≥ 10 mm with spiral CT or MRI
   * Bone lesions: lytic or mixed (lytic + sclerotic) in the absence of measurable disease as defined above.
6. Adequate bone marrow and coagulation according RCP
7. Adequate liver function, according RCP
8. Adequate renal function, according RCP
9. ECOG Performance Status ≤ 2
10. Written informed consent

Exclusion Criteria:

1. HER2-overexpressing patients by local laboratory testing (IHC3+ staining or in situ hybridization positive).
2. Patients who received chemotherapy for MBC
3. Patients who received more than one NSAI treatment for LABC or MBC
4. Pre-menopausal, pregnant, lactating women.
5. Known hypersensitivity to mTOR inhibitors
6. Patients with rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose galactose malabsorption.
7. Radiotherapy within four weeks prior to enrollment
8. Currently receiving hormone replacement therapy, unless discontinued prior to enrollment.
9. Patients receiving concomitant immunosuppressive agents or chronic corticosteroids use, at the time of study entry except in some cases
10. Patients with symptomatic visceral disease in need of urgent disease control
11. Symptomatic brain or other CNS metastases.
12. Patients with a known history of HIV seropositivity.
13. Active, bleeding diathesis, or on oral anti-vitamin K medication (except cases).
14. Any severe and / or uncontrolled medical conditions such as:

    * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to enrollment, serious uncontrolled cardiac arrhythmia
    * Uncontrolled diabetes as defined by fasting serum glucose > 1.5 × ULN
    * Acute and chronic, active infectious disorders
    * Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the study treatments (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome)
    * Inability to swallow oral medications
    * Significant symptomatic deterioration of lung function.
15. Hepatic-related exclusion criteria:

    * History of liver disease, such as cirrhosis or chronic active hepatitis B and C.
    * Presence of Hepatitis B surface antigen (HbsAg) and/or of Hepatitis B Virus - Deoxyribonucleic acid (HBV-DNA)
    * Presence of anti-HCV and/or HCV-RNA-PCR
    * History of, or current alcohol misuse/abuse within the past 12 months
    * Patients being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A within the last 5 days prior to enrollment.
    * History of non-compliance to medical regimens.
    * Patients unwilling to or unable to comply with the protocol
16. Patients being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A
17. History of non-compliance to medical regimens.
18. Patients unwilling to or unable to comply with the protocol.

Screening for hepatitis B

Prior to enrollment, peculiar patients should be tested for hepatitis B viral load and serologic markers, that is, HBV-DNA, HBsAg, HBsAb, and HBcAb:

Screening for hepatitis C Patients with any of the following risk factors for hepatitis C should be tested

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 745 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS1) | Time elapsed from randomization to progression or death for any cause whichever occurred first assessed up to 30 months
  The number of events required for the other primary endpoint (PFS1), and the expected time needed to achieve it are derived from previous calculations. Assuming an average accrual rate of 31 pts/month (677pts/22 months), a median PFS1 of 6 months in the Fulvestrant arm (control), a Hazard ratio of 0.70 (implying that a median PFS1 of 8,6 months is expected in the experimental arm, a 2-sided significance level of 0.025 and power of 0.90, 391 events are required for PFS1, that will be achieved in about 22 months (East 6 software).
Total Progression-free survival (PFST) | Time elapsed from randomization to progression or death for any cause whichever occurred first assessed up to 30 months
  Overall study size is driven by the endpoint less frequent (PFST). Sample size is planned to identify a Hazard ratio of 0.75, assuming an overall study duration of 36 months, an accrual duration of 24 months, a 2-sided significance level of 0.025 and power of 0.80. Assuming a median PFST of 12 months in the Fulvestrant arm (control), the expected PFST in the experimental arm will be equal to 16 months and 677 subjects need to be enrolled (East 6 software) with an average accrual rate equal to 30.8 patients/month (11 months per year have been considered).

SECONDARY OUTCOMES:
Response Rate | Time elapsed from randomization to progression or death for any cause whichever occurred first assessed up to 30 months
  Objective Response Rate (ORR), the Clinical Benefit, the overall survival, and the safety profile and the QOLof of the sequence of fulvestrant followed, at progression by exemestane and everolimus versus the sequence of examestane and everolimus followed, at progression, by fulvestrant in postmenopausal women with HR + and HER2- LABC or MBC previously treated with NSAI in the adjuvant or metastatic setting.
Clinical Benefit Rate | Time elapsed from randomization to progression or death for any cause whichever occurred first assessed up to 30 months
  Objective Response Rate (ORR), the Clinical Benefit, the overall survival, and the safety profile and the QOLof of the sequence of fulvestrant followed, at progression by exemestane and everolimus versus the sequence of examestane and everolimus followed, at progression, by fulvestrant in postmenopausal women with HR + and HER2- LABC or MBC previously treated with NSAI in the adjuvant or metastatic setting.
Overall Survival | Time elapsed from randomization to progression or death for any cause whichever occurred first assessed up to 30 months
  Objective Response Rate (ORR), the Clinical Benefit, the overall survival, and the safety profile and the QOLof of the sequence of fulvestrant followed, at progression by exemestane and everolimus versus the sequence of examestane and everolimus followed, at progression, by fulvestrant in postmenopausal women with HR + and HER2- LABC or MBC previously treated with NSAI in the adjuvant or metastatic setting.
Safety - 5D5L questionnaire | up to 31 days since last treatment
  The overall observation period will be divided into three mutually exclusive segments per treatment phase:
  1. pre-treatment period: from day of patient's informed consent to the day before first dose of study medication (phase 1) on-treatment period: from day of first dose of study medication to 30 days (minimum washout) after last dose of study medication (phase 2) or first dose of second phase treatment after cross-over
  2. post-treatment period: starting at day 31 after last dose of study medication (phase 2)

CONTACTS AND LOCATIONS:
Overall Officials: Sabino De Placido, MD, Principal Investigator — Dipartimento di Medicina Clinica e Chirurgia Oncologia Università degli Studi di Napoli "Federico II"
Locations (41):
- Italy (41):
  - ASL19 - Ospedale Cardinal Massaia, Asti
  - Azienda Ospedaliera Policlinico di Bari, Bari
  - Istituto Tumori Giovanni Paolo II, Bari
  - Azienda Ospedaliera "G. Rummo", Benevento
  - Ospedale Fatebenefratelli 'Sacro Cuore di Gesù' di Benevento, Benevento
  - A.O. Ospedale Papa Giovanni XXIII, Bergamo
  - Presidio Ospedaliero Antonio Perrino, Brindisi
  - Azienda Ospedaliera - A. Businco - A.S.L. N. 8, Cagliari
  - Fondazione del Piemonte per l' Oncologia - Istituto di Ricovero e Cura a Carattere Scientifico (I.R.C.C.S.), Candiolo
  - ASL di Taranto - Polo Occidentale, Castellaneta
  - A.O.R.N.A.S. Garibaldi Nesima di Catania, Catania
  - Fondazione per la Ricerca e la Cura dei Tumori T. Campanella - Campus S. Venuta, Catanzaro
  - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - Ospedale Infermi di Rimini, Faenza
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Ospedaliero - Universitaria Ospedali Riuniti di Foggia, Foggia
  - I.R.C.C.S. A.O.U San Martino - IST, Genova
  - Ospedale Civile di guastalla, Guastalla
  - Presidio Ospedaliero "Renzetti", Lanciano
  - Ospedale Vito Fazzi, Lecce
  - Ospedale Civile San Salvatore - Università degli Studi L'Aquila, L’Aquila
  - Ospedale di Macerata, Macerata
  - AO Papardo, Messina
  - AORN . Ospedali dei colli Monaldi-Cotugno, Napoli
  - Azienda Ospedaliera 'A. Cardarelli' (AORN), Napoli
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Istituto Nazionale per lo studio dei Tumori - Fondazione 'Pascale', Napoli
  - A.O.U. 'Maggiore della Carità', Novara
  - A.O.U.P. 'Paolo Giaccone', Palermo
  - Azienda Ospedaliera S. Chiara, Pisa
  - Ospedale F. Lotti, Pontedera
  - Ospedale di Ravenna, Ravenna
  - Campus Biomedico di Roma, Roma
  - Istituto Regina Elena per lo studio e la cura dei tumori - Oncologia A, Roma
  - Istituto Regina Elena per lo studio e la cura dei tumori - Oncologia B, Roma
  - Azienda Ospedaliera 'San Giovanni di Dio e Ruggi D'Aragona', Salerno
  - IRCCS - Istituto di Ricovero e Cura a Carattere Scientifico 'Casa Sollievo della Sofferenza', San Giovanni Rotondo
  - Azienda Ospedaliera Universitaria di Sassari, Sassari
  - Azienda Ospedaliero Universitaria ´S. Maria della Misericordia´ di Udine, Udine
  - "Ospedale Borgo Roma Verona Sezione di Oncologia Medica", Verona
  - Ospedale Sacro Cuore Don Calabria di Negrar, Verona

IPD SHARING:
Plan to Share IPD: No